CLINICAL TRIAL: NCT05535452
Title: Photobiomodulation for Prevention of Radiodermatitis in Women With Breast Cancer Undergoing Adjuvant Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Principal Investigator, Rejane Medeiros Costa, Physiotherapist, Instituto Nacional de Cancer, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Prevention of radiodermatitis
Record Dates: First submitted 2022-08-24; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Radiodermatitis
Keywords: radiotherapy; Radiodermatitis; photobiomodulation; breast cancer
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: After recruitment, the women will be allocated to: Intervention Group and Control Group. The randomization of the study will be performed in an allocation ratio of 1:1 for the two groups and generated per block of envelopes, sealed and opaque, every 10 patients, which will contain the allocation code (five codes for the intervention group and five codes for the control group). This choice was chosen to avoid influences of the therapist's or patient's preference in relation to the intervention. The patients will be oriented in relation to the group that will be inserted and that the follow-up will be performed while the patient is on radiotherapy and up to three months after treatment. All evaluations, intervention and data collection will be performed by professionals trained and qualified for this purpose.
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the nature of the intervention, physiotherapists who supervise the application of the photobiomodulation technique will not be blinded and only patients and evaluators of the results will be blinded to the allocation of the groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group control (Placebo Comparator): Patients will receive applications with the LED board turned off without light activation. Applications will be performed within 1 hour after radiotherapy, three times a week, by a trained team, consisting of physical therapists and physical therapy students, and the application time will be the same as in the intervention group. Women will be instructed to maintain specific home exercises for the upper limbs, which are part of the routine of the physiotherapy sector since the first postoperative day at the HCIII/INCA, in addition to their usual physical activities.
  Interventions: Device: Photobiomodulation through LED board
- Intervention group (Experimental): At the beginning of radiotherapy treatment, all HCIII/INCA patients are instructed by the nursing team in this sector to use the DNA® ointment provided at the institution and to take proper skin care. Patients identified by the nursing staff with some degree of radiodermatitis undergo treatment with silver sulfadiazine and, if necessary, radiotherapy can be interrupted so that the skin regenerates.
  Interventions: Device: Photobiomodulation through LED board

INTERVENTIONS:
Device: Photobiomodulation through LED board — The applications will be performed within 1 hour after radiotherapy, three times a week, by a trained team, consisting of physiotherapists and physiotherapy students, through the sportllux LED plate equipment, medium size, which combines light emitters in two wavelengths: red (660nm) and infrared (850nm).
  Other Names: Light emitting diode

SUMMARY:
This is a Randomized Controlled Clinical Trial Women with breast cancer who are indicated for treatment with adjuvant radiotherapy will be eligible. Patients who underwent surgery and/or chemotherapy outside the institution and patients with comprehension difficulties will be excluded. After recruitment, women will be allocated into two groups: intervention (use of LED board) and control (placebo board). The degree of radiodermatitis, pain, edema and/or lymphedema, paresthesia, functionality, quality of life, skin conditions and related independent variables, such as the characteristics of the patient, the tumor and the oncological treatment performed will be evaluated. Thus, the hypothesis of the study is the prevention of radiodermatitis, which is a complication of radiotherapy treatment using photobiomodulation with LED board as a means of intervention.

DETAILED DESCRIPTION:
Introduction: For Brazil, the INCA estimate is 66,280 new cases of breast cancer for each year of the 2020-2022 triennium. The treatment of breast cancer depends on the stage of the disease and the type of tumor. Treatment modalities are divided into systemic (chemotherapy, hormone therapy and biological therapy) and local (radiotherapy and surgery) that can be performed alone or in combination, according to clinical and tumor characteristics. Radiotherapy is associated with some adverse effects, including radiodermatitis, which is characterized by tissue damage that occurs immediately after the first radiotherapy session and, as subsequent sessions occur, resulting from dose fractionation, it starts to the dose accumulates in the skin, which causes the recruitment of inflammatory cells and the worsening of this complication. General objective: To evaluate the effectiveness of photobiomodulation with the application of the LED board in the prevention of radiodermatitis in women with breast cancer undergoing adjuvant radiotherapy at the Cancer Hospital III of the National Cancer Institute (HCIII/INCA). Materials and methods: This is a Randomized Controlled Clinical Trial Women with breast cancer who are indicated for treatment with adjuvant radiotherapy will be eligible. Patients who underwent surgery and/or chemotherapy outside the institution and patients with comprehension difficulties will be excluded. After recruitment, women will be allocated into two groups: intervention (use of LED board) and control (placebo board). The degree of radiodermatitis, pain, edema and/or lymphedema, paresthesia, functionality, quality of life, skin conditions and related independent variables, such as the characteristics of the patient, the tumor and the oncological treatment performed will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age
* Stage I to IIIC breast cancer
* Have an indication for adjuvant radiotherapy treatment at HCIII/INCA.

Exclusion Criteria:

* have a previous diagnosis of cancer
* underwent surgery and/or chemotherapy outside the Institution
* were unable to respond to the questionnaires
* were unable to receive photobiomodulation due to acute infections will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women diagnosed with breast cancer and indicated for adjuvant radiotherapy
Enrollment: 148 (Estimated)
Dates: Start 2023-02-06 (Estimated); Primary Completion 2024-02-06 (Estimated); Study Completion 2025-02-06 (Estimated)

PRIMARY OUTCOMES:
Degree of Radiodermatitis | one day, 30 days, 3 and 6 months after radiotherapy treatment
  Objective scoring of the severity of radiodermatitis using the classification system of the Radiotherapy Oncology Group / European Organization for Research and Treatment of Cancer (RTOG / EORTC), where the set of skin reactions caused by radiotherapy is classified as grade 0: when there is no reaction; grade 1: mild erythema, epilation and dry flaking; grade 2: painful erythema, moist flaking, and moderate edema; grade 3: wet flaking, confluent and important edema; ulceration, bleeding and necrosis.

SECONDARY OUTCOMES:
Pain at the application site | one day, 30 days, 3 and 6 months after radiotherapy treatment
  Pain - pain assessment using the visual analog scale (VAS). Pain will be assessed weekly by the patient. Patients will respond to the visual analog scale modified for pain (self-assessment of the patient).
Edema/Lymphedema | one day, 30 days, 3 and 6 months after radiotherapy treatment
  Edema/Lymphedema: Edema or lymphedema in the upper limb homolateral to axillary breast cancer surgery will be evaluated by perimetry in the upper limbs. The points of the measurements will be: elbow joint interline (IAC), 07 cm above the IAC, 14 cm above the IAC, 7 cm below the IAC, 14 cm below the IAC, 21 cm below the IAC and back of the hand. The total volume of the limb will be calculated by the cone trunk formula, using the circumference measurements:
  V = h * (C² + Cc + c²) / (- * 12). Where, V is the total volume, C and c are the circumferences between the measured points and h is the distance between the circumferences in each segment. Lymphedema will be considered when the total volume is 200 ml between the affected limb and the contralateral limb, 6 months after surgical treatment. Edema will be considered when the total volume is 200 ml in the first six months after surgery.
Paresthesia | one day, 30 days, 3 and 6 months after radiotherapy treatment
  It can be evaluated using the Stesiometer (monofilaments) . Patients will be evaluated in a quiet and comfortable environment with as little interference as possible; will face the examiner with the hand or foot supported; the test will be demonstrated to the patient using an area of skin with normal sensitivity; patients will be blinded or instructed to close their eyes; the test will start following the specific technique according to the instrument used; the points tested will be previously determined. The testing sequence can be random.
Functionality | one day, 30 days, 3 and 6 months after radiotherapy treatment
  DASH Questionnaire. This questionnaire is about symptoms as well as skills to do certain activities. Must be answered with regards to last week's physical condition. If you were unable to perform physical activity in the past week, estimate which answer would be correct. It doesn't matter which hand or arm is used to do the activity, the response is based on skill regardless of how the task is performed. It has 30 questions and two optional modules and uses a 5-point scale and the total score ranges from 0 (no dysfunction) to 100 (severe dysfunction).
Skin quality | one day, 30 days, 3 and 6 months after radiotherapy treatment
  Skindex: Questionnaire used to evaluate patients with any skin alteration and allows identifying how they evolve over time after treatment. In this scale, responses are reported on 3 scales or dimensions: physical (items number 1 to 4), emotions (items number 5 to 11) and functionality (items number 12 to 16). Responses are given on a 7-point Likert-type scale, ranging from 0 ("never bothered") to 6 ("always bothered"), according to the intensity of the frequency with which the patient was bothered, due to his skin condition during the last seven days. All responses are transformed into a linear scale ranging from 0 to 100. The scores for each of the 3 domains (symptoms, emotions and functionality) are calculated. The higher the value found, the worse the quality of life.
Questionnaire about Health-related quality of life | one day, 30 days, 3 and 6 months after radiotherapy treatment
  will be the EORTC QLQ-C30 3rd version, translated into Portuguese, multidimensional and self-administered, which includes 30 questions related to five functional scales (physical, functional, emotional, social and cognitive), a scale on health status assessment, three symptom scales (fatigue, pain, and nausea/vomiting) and six additional symptom items (dyspnea, insomnia, loss of appetite, constipation, diarrhea, and financial difficulties). And the specific quality of life questionnaire for breast cancer patients, the EORTC QLQ-BR23, translated into Portuguese, which contains 23 questions related to a functional scale (body image, sexual function, sexual pleasure and future perspectives) and a scale of symptoms (side effects of systemic therapy, breast symptoms, arm symptoms and hair loss). Both questionnaires will be applied in relation to the last week of the patient and both were translated and validated into Portuguese.
Questionnaire about Satisfaction with photobiomodulation | one day, 30 days, 3 and 6 months after radiotherapy treatment
  Self-report on efficacy and overall satisfaction with the management of radiodermatitis.
Questionnaire about Impact of radiodermatitis | one day, 30 days, 3 and 6 months after radiotherapy treatment
  Self-report on the impact of radiodermatitis on activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Rejane M Costa, PhD, Principal Investigator — National Cancer Institute - INCA

IPD SHARING:
Plan to Share IPD: No